CLINICAL TRIAL: NCT00934622
Title: Visual Function After Implantation of Bilateral AcrySoft ReSTOR Aspheric Intraocular Lens (IOL)
Brief Title: Visual Function After Implantation of Bilateral AcrySoft ReSTOR Aspheric IOL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Doug Hubatsch\Clinical Research Director, Alcon Research
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALCONsur002.07
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Results first posted 2010-05-06 (Estimated); Last update posted 2010-05-06 (Estimated); Status verified 2010-05

CONDITIONS: Cataract
Keywords: AcrySof; ReSTOR; Aspheric IOL; Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AcrySof® ReSTOR® Aspheric IOL (Experimental): AcrySof® ReSTOR® Aspheric Intraocular Lens (IOL)
  Interventions: Device: AcrySof® ReSTOR® Aspheric IOL

INTERVENTIONS:
Device: AcrySof® ReSTOR® Aspheric IOL — AcrySof® ReSTOR® Aspheric Intraocular Lens (IOL) implanted into the study eye following the cataract extraction surgery

SUMMARY:
This study will involve up to 20 bilateral patients per surgeon. Patients will be assessed pre-operatively, and at subsequent visits (following the implantation of the intraocular lens in the second eye) at 1 week, 1 month, 3 months and 6 months post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* 21 years or older;
* need spherical correction between 10-30 Diopters (D);
* corneal astigmatism less than 0.75D as measured by keratometry;
* willing to sign an Informed Consent Form and complete all visits;
* pupil dilation greater than 6mm;
* expected Visual Acuity (measured in logMAR)=0.3 or better

Exclusion Criteria:

* Women of childbearing potential;
* irregular corneal astigmatism;
* keratopathy/keratectasia;
* cornea inflammation or edema;
* cornea reshaping surgery;
* corneal dystrophy;corneal transplant;
* amblyopia;
* glaucoma;
* Retinal Pigment Epitheliopathy (RPE)/Macular changes;
* proliferative diabetic retinopathy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2007-11; Primary Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects >21 years of age, either sex, and any race. Diagnosis of cataracts in both eyes. 27-Jun-2007 to 20-May-2009
Pre-assignment Details: Subject's eligibility was determined at the preoperative visit. All subjects met inclusion/exclusion criteria.
Period: Overall Study
Arm/Group | AcrySof® ReSTOR® Aspheric IOL
Started | 76
Completed | 68
Not Completed | 8
Not completed — Lost to Follow-up | 7
Not completed — 2nd Intraoperative exclusion criteria | 1

BASELINE CHARACTERISTICS:
Arm/Group | AcrySof® ReSTOR® Aspheric IOL
Number analyzed (Participants) | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 43
Gender [Number; unit: participants] — Gender data not collected for 1 patient.
  participants
    Female | 48
    Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: Comparison of visual acuity (measured in logMAR) prior to and following bilateral implantation of the AcrySof ReSTOR Aspheric Intraocular Lens (IOL). Visual parameters were assessed prior to and after the implantation of the second lens at 1 week, 1 month, 3 months, and 6 months. LogMAR, the unit of measure for visual acuity, is the "logarithm of the minimum angle of resolution". A lower logMAR value indicates better visual acuity.
Time Frame: pre-operative;1 week,1 month, 3 months and 6 months after 2nd eye surgery
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | AcrySof® ReSTOR® Aspheric IOL
Number analyzed (Participants) | 76
logMAR
  Preoperative | 0.54 (0.3)
  1 Week | 0.06 (0.12)
  1 Month | 0.03 (0.08)
  3 Months | 0.04 (0.08)
  6 Months | 0.05 (0.09)

2. Secondary Outcome: Spectacle Independence
Description: Spectacle independence is the percentage of patients that do not always need to wear glasses. This outcome measure is patient reported.
Time Frame: pre-op;1 week,1 month,3 months and 6 months after 2nd eye surgery
Population: Patient population was not consistent throughout the study. Number of patients analyzed at each visit is as follows: Preoperative n=76, Week 1 n=61, 1 Month n=71, 3 Months n=70, 6 Months n=68.
Measure: Number; unit: Percentage of Participants
Arm/Group | AcrySof® ReSTOR® Aspheric IOL
Number analyzed (Participants) | 76
Percentage of Participants
  Preoperative | 29
  1 Week Postoperative | 96.8
  1 Month Postoperative | 97.2
  3 Months Postoperative | 98.6
  6 Months Postoperative | 100

ADVERSE EVENTS:
Time Frame: June 27, 2007 (First Subject, first visit) through August 1, 2009 (Last subject, last visit)
Arm/Group | AcrySof® ReSTOR® Aspheric IOL
Serious Adverse Events (participants affected / at risk) | 0/76
Other Adverse Events (participants affected / at risk) | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less